CLINICAL TRIAL: NCT06649552
Title: French Validation of Schizophrenia Proneness Instrument- Child Youth
Acronym: SPI-CY-Fr
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A01301-46
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Clinical High Risk for Psychosis (CHR)
Keywords: SPI-CY; Basic Symptoms; Psychosis; Clinical High Risk; Ultra High Risk
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPI-CY assessment (Other): all patients will undergo a SPI-CY interview
  Interventions: Diagnostic Test: Psychiatric and psychological diagnostic tests

INTERVENTIONS:
Diagnostic Test: Psychiatric and psychological diagnostic tests — French validation of the SPI-CY

SUMMARY:
The clinical concept of a at risk mental state of developing psychosis is based on the identification of attenuated psychotic symptoms during the prodromal phase of psychoses (Schmidt et al., 2015). Early detection and support of these symptoms can delay the risk of transition to a first psychotic episode (van der Gaag, van den Berg, & Ising, 2019).

The Basic Symptom approach enables detection at the earliest stage of the prodromal phase. It postulates that subtle, subjective manifestations predating attenuated psychotic symptoms are present very early in the prodromal phase of psychosis and also have predictive value for the risk of developing psychosis (F. Schultze-Lutter, 2009). Basic symptoms are assessed using the Schizophrenia Proneness Instrument, available in an adult (SPI-A) and child/adolescent (SPI-CY) version. These scales are part of the international recommendations for the assessment of patients with a Clinical State at High Risk of Psychosis (CHR-P) (Schmidt et al., 2015; F Schultze-Lutter et al., 2015). The SPI-A is validated in French under the name "Outil d'Evaluation du Risque Schizophrénique version adulte (OERS-A)" (Schultze-Lutter et al., 2007. French translation by JR. Teyssier with the collaboration of F. Gamma and P. Loulergue), but no French version of the SPI-CY has yet been validated.

In collaboration with Dr. Frauke Schultze-Lutter, the investigators have recently published a French translation of the SPI-CY (Schizophrenia Predisposition Instrument - Version for Children and Adolescents, F. Schultze-Lutter, M. Marshall, E. Koch, 2021. French translation by F. Bernardin and C. Dondé). This French translation must now be validated to ensure the inter-rater fidelity of the interview.

We therefore propose to study the inter-rater reliability of the French version of the SPI-CY by comparing ratings between clinicians who have undergone training in basic symptoms and in administering the SPI-A and SPI-CY tools by Dr. Schultze-Lutter. This validation will be carried out by comparing, on the one hand, the rating of the SPI-CY by a clinician A who has administered it to the patient and, on the other hand, the blind rating of a clinician B on the basis of the interview recorded by clinician A with his patient.

The investigators will also explore the links between the SPI-CY and other clinical scales such as the Multisensory Hallucination SCale (MHASC) (Demeulemeester et al., 2015), the Prodromal Questionnaire 16 (PQ-16) (Lejuste et al., 2021), the Audiograph (Giersch, Huard, Park, & Rosen, 2021) and the Perceptual and Cognitive Aberrations (PCA) (McDonald et al., 2019).

ELIGIBILITY:
Inclusion Criteria :

* Patients (men or women) followed at one of the 3 following structures in France : CLIP-Ado Nancy, CH Alpes-Isère, CHRU Lille for a suspected mental state at risk of developing psychosis, as determined by the CAARMS scale and/or the SPI-CY scale.
* Age between 12 and 17 years and 11 months
* Affiliation with a social security scheme or beneficiary of such a scheme.
* Native language: French.
* Adolescents who have been informed of the study, have received the study information note and have not objected to participating in the study
* At least one of the holders of parental authority having been informed of the study, having received the relevant information note and not having objected to the adolescent participation
* Consent to audio recording of the SPI-CY scale administration: for the adolescent and at least one parent.

Exclusion Criteria:

* Pregnant woman, parturient or nursing mother
* Person deprived of liberty by judicial or administrative decision
* Person in a life-threatening emergency
* Impairment of the subject that makes it difficult, if not impossible, to participate in the trial or to understand the information provided.
* Abuse or dependence on any substance according to DSM V criteria, excluding cannabis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
SPI-CY assessment : Schizophrenia Proneness Instrument - Child and Youth version | Day 1

SECONDARY OUTCOMES:
CAARMS assessment : Comprehensive Assessment of At Risk Mental State | Day 15 maximum
MHASC assessment : Multisensory HAllucination SCale | Day 15 maximum
PQ16 assessment : Prodromal Questionnaire 16 | Day 15 maximum
PCA assessment : Perceptual and Cognitive Aberrations | Day 15 maximum
Audiograph : formalization of visual hallucinations | Day 15 maximum

CONTACTS AND LOCATIONS:
Overall Officials: Florent BERNARDIN, Principal Investigator — Centre Psychothérapique de Nancy (CPN)
Locations (3):
- France (3):
  - CHRU Lille, Lille
  - Centre Psychothérapique de Nancy, Nancy
  - CH Alpes-Isère, Saint-Egrève

IPD SHARING:
Plan to Share IPD: Yes